CLINICAL TRIAL: NCT03999775
Title: Effect on Bone Biomarkers and Bone Mineral Density and Tolerability of Calcium and Vitamin D Supplementation With and Without Collagen Peptides in Postmenopausal Women With Osteopenia
Brief Title: Effect of Calcium and Vitamin D Supplementation With and Without Collagen Peptides in Postmenopausal Women With Osteopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ioannis K. Triantafyllopoulos, MD,MSci,PhD (Other)
Responsible Party: Sponsor-Investigator, Ioannis K. Triantafyllopoulos, MD,MSci,PhD, Assistant Professor of Orthopaedics, National and Kapodistrian University of Athens
Organization: National and Kapodistrian University of Athens (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 84908/2017
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Osteopenia; Postmenopausal Osteopenia
Keywords: Collagen peptides; Bone turnover markers; Calcium supplement; Postmenopausal women
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Calcium; Vitamin D

ARMS (2):
- Calcium, vitamin D and bioactive collagen peptides supplement (Active Comparator): In this arm, all patients received a sachet containing 5mg bioactive collagen peptides, 500 mg calcium lactate and 400 IU vitamin D3 per day.
  Interventions: Dietary Supplement: Calcium, vitamin D and bioactive collagen peptides supplement
- Calcium and vitamin D supplement (Active Comparator): In this arm, all patients received a chewable tablet containing 500 mg calcium carbonate and 400 IU vitamin D3 per day.
  Interventions: Dietary Supplement: Calcium and vitamin D supplement

INTERVENTIONS:
Dietary Supplement: Calcium, vitamin D and bioactive collagen peptides supplement
  Arms: Calcium, vitamin D and bioactive collagen peptides supplement
Dietary Supplement: Calcium and vitamin D supplement
  Arms: Calcium and vitamin D supplement

SUMMARY:
Osteoporosis is undoubtedly one of the most common diseases affecting older individuals with debilitating consequences. Osteopenia, defined as T-score between -1 and -2.5, has also been associated with increased risk of osteoporotic fractures and the associated morbidity and mortality. Prompt diagnosis, prevention and treatment of both osteopenia and osteoporosis are essential in order to minimize future fracture risk. The mainstay of treatment of osteopenia and osteoporosis includes dietary changes, regular weight-bearing exercises, calcium and vitamin D supplementation and pharmacologic treatment mainly with antiresorptive or anabolic agents. Collagen peptides (CPs), also called collagen hydrolysates produced by hydrolysis of collagen, have also been shown to have high oral bioavailability and could have a place as a treatment option.

Type I collagen comprises approximately 95% of the entire collagen content of bone. Bone matrix, unlike other connective tissues, possesses the unique ability to become calcified. Spindle or plate-shaped crystals of hydroxyapatite are found between and around collagen fibers, oriented in the same direction as collagen fibers are. Nowadays, it is well-documented that type I collagen molecules are involved in the mechanical properties of bone. Collagen peptide compounds seem to exert their beneficial effect on bone by affecting bone remodeling and mineralization of the bone matrix, promoting the proliferation and differentiation of pre-osteoblasts while reducing the maturation of osteoclasts. Several preclinical studies performed in mice and rats support this notion and also suggested that orally administrated CPs increased bone mineral density (BMD), as well as the compositional and the biodynamic characteristics of vertebrae. Human studies in postmenopausal women have also yielded positive results with increased BMD and blood biomarkers after 6 months and 1 year of oral administration.

The aim of the present randomized prospective study was to examine and compare the efficacy, as represented by the changes in bone biomarkers procollagen type I N-terminal propeptide (P1NP) and C-terminal telopeptide of collagen I (CTX), and bone mineral density and the tolerability of supplementation of calcium, vitamin D with and without bioactive CPs for a year in postmenopausal women with osteopenia.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* T-score in the osteopenic range (-1.0 > T-score > -2.5) at either the lumbar spine (LS) or femur as measured by dual energy X-ray absorptiometry (DXA)

Exclusion Criteria:

* T-score in the osteoporotic range (T-score < -2.5) at any site
* Patients receiving supplements of calcium and/or vitamin D at that time or during the last year
* Patients receiving medications known to positively or negatively affect bone turnover or BMD at that time or during the last 3 years (e.g. antiresorptive agents, oestrogens, systemic corticosteroids), or
* Secondary cause of osteoporosis (e.g. alcohol abuse, thyrotoxicosis etc)
* Patients who did not attend to their follow-up appointment and consequently had only the baseline measurements

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Postmenopausal osteopenia
Enrollment: 51 (Actual)
Dates: Start 2017-01-14 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Comparison of %-changes of P1NP and CTX levels from baseline to 3 months of supplementation between the two groups. | 3 months
  The primary endpoint of the study was the comparison of %-changes of P1NP and CTX levels from baseline to 3 months of supplementation between the two groups.

SECONDARY OUTCOMES:
Change of P1NP and CTX levels within groups and comparison of the adverse effects (tolerability), and/or the adherence to treatment between the two groups. | 3 months
  The secondary endpoints were the change of P1NP and CTX levels following the 3-month calcium and vitamin D supplementation with and without collagen peptides supplement, the comparison of adverse effects (tolerability), and/or the adherence to treatment between the two groups.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Argyrou C, Karlafti E, Lampropoulou-Adamidou K, Tournis S, Makris K, Trovas G, Dontas I, Triantafyllopoulos IK. Effect of calcium and vitamin D supplementation with and without collagen peptides on bone turnover in postmenopausal women with osteopenia. J Musculoskelet Neuronal Interact. 2020 Mar 3;20(1):12-17. PMID 32131366